CLINICAL TRIAL: NCT03616964
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study of Baricitinib in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of Baricitinib in Participants With Systemic Lupus Erythematosus (SLE-BRAVE II)
Acronym: BRAVE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16677; I4V-MC-JAIA (Other: Eli Lilly and Company); 2017-005027-25 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 milligram (mg) Baricitinib (Experimental): Participants received one 2 mg baricitinib tablet and one placebo tablet matching 4 mg baricitinib administered orally once daily (QD) for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 4 mg Baricitinib (Experimental): Participants received one 4 mg baricitinib tablet and one placebo tablet matching 2 mg baricitinib administered orally QD for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Participants received 2 placebo tablets: one placebo tablet matching 4 mg baricitinib and one placebo tablet matching 2 mg baricitinib administered orally QD for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 2 milligram (mg) Baricitinib; 4 mg Baricitinib
Drug: Placebo — Administered orally

SUMMARY:
The reason for this study is to see how effective and safe the study drug known as baricitinib is in participants with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of SLE at least 24 weeks prior to screening.
* Have documentation of having met at least 4 of 11 Revised Criteria for Classification of Systemic Lupus Erythematosus according to the 1997 Update of the 1982 American College of Rheumatology (ACR) criteria for classification of SLE prior to randomization.
* Have a positive antinuclear antibody (ANA) (titer ≥1:80) and/or a positive anti-double-stranded deoxyribonucleic acid (dsDNA), and/or a positive anti-Smith (anti-Sm) as assessed by a central laboratory during screening.
* Have a total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥6 during screening.
* Have a clinical SLEDAI-2K score ≥4 at randomization.
* Have at least 1 British Isles Lupus Assessment Group (BILAG) A score or 2 BILAG B scores during screening.
* Are receiving at least one of the following standard of care medications for SLE:

  * A single antimalarial at a stable dose for at least 8 weeks prior to screening
  * A single immunosuppressant at a stable dose for at least 8 weeks prior to screening
  * An oral corticosteroid, initiated at least 4 weeks prior to screening, at a stable dose ≤40 milligrams/day prednisone (or equivalent) for at least 2 weeks prior to screening. If the participant is not receiving an antimalarial or immunosuppressant, the dose of corticosteroid must be ≥7.5 milligrams/day prednisone (or equivalent)

Exclusion Criteria:

* Have severe active lupus nephritis.
* Have active central nervous system (CNS) lupus.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection.
* Have received cyclophosphamide (or any other cytotoxic agent) within 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (159):
- United States (39):
  - University of Arizona Arthritis Center, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Tucson, Arizona
  - Wallace Rheumatic Studies Center, Beverly Hills, California
  - Medvin Clinical Research - Weidmann, Covina, California
  - Office: Dr Robin K Dore, Tustin, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Millennium Research, Ormond Beach, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - North Georgia Rheumatology, PC, Lawrenceville, Georgia
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Advanced Rheumatology, PC, Lansing, Michigan
  - Glacier View Research Institute - Endocrinology, Kalispell, Montana
  - Innovative Health Research, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Arthritis and Osteoporosis Associates of New Mexico, Las Cruces, New Mexico
  - St. Lawrence Health System, Canton, New York
  - New York University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Joint and Muscle Medical Care, Charlotte, North Carolina
  - Box Arthritis & Rheumatology of the Carolinas, PLLC, Charlotte, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Articularis Healthcare d/b/a/ Low Country Rheumatology, PA, Summerville, South Carolina
  - Eagle Medical, Crossville, Tennessee
  - Dr. Dhiman Basu Private Practice, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - Clear Lake Specialties, Webster, Texas
  - Arthritis Clinic of Northern VA, P.C., Arlington, Virginia
  - Spectrum Medical Inc., Danville, Virginia
- Argentina (11):
  - Aprillus Asistencia e Investigacion - Servicio de neurologia, CABA, Buenos Aires
  - DOM Centro de Reumatologia, Ciudad de Buenos Aires, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Comite de Etica en Investigacion - CEMIC, Buenos Aires, Ciudad Autonoma de Buenos Aire
  - Clinica Adventista Belgrano, CABA, Ciudad Autónoma de Buenos Aire
  - Sanatorio Británico, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman, Tucumán Province
  - Sanatorio Guemes Cardiocirugia, Ciudad Autonoma Buenos Aires
  - IR Medical Center S.A. Instituto de Reumatologia, Mendoza
- Chile (6):
  - Clinical Research Chile SpA, Valdivia, Los Ríos Region
  - Enroll SpA, Providencia, Región Metropolitana de Santia
  - Clinica Alemana de Osorno, Osorno
  - Sociedad Medica Del Aparato Locomotor SA, Santiago
  - Prosalud y cia. Ltda., Santiago
  - ReumaCen Centro Reumatologico Integral, Viña del Mar
- Colombia (8):
  - HPTU-El Hospital con alma Pablo Tobon Uribe, Medellín, Antioquia
  - Circaribe SAS, Barranquilla, Atlántico
  - Clinica de la Costa, Barranquilla, Atlántico
  - Idearg S.A.S., Bogota, Cundinamarca
  - Centro Integral de Reumatologia e Inmunologia, Bogotá, Cundinamarca
  - Servimed S.A.S., Bucaramanga, Santander Department
  - Centro de Medicina Interna, Cali, Valle del Cauca Department
  - Preventive Care Ltdac, Chía
- France (5):
  - CHRU Brest - Hopital Cavale Blanche, Brest, Finistère
  - Centre hospitalier universitaire de Haut Leveque, Pessac, Gironde
  - CHU Montpellier Lapeyronie Hospital, Montpellier, Hérault
  - Centre hospitalier universitaire Pellegrin, Bordeaux
  - Hopital Européen, Marseille
- India (14):
  - Krishna Institute of Medical Science, Hyderabad, Andhra Pradesh
  - Panchshil Hospital, Ahmedabad, Gujarat
  - CIMS Hospital Private Limited, Ahmedabad, Gujarat
  - NHL Municipal Medical College & VS General Hospital, Ahmedabad, Gujarat
  - Shree Giriraj Hospital, Rajkot, Gujarat
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Sterling Hospital, Vadodara, Gujarat
  - St. John Medical College & Hospital, Bangalore, Karnataka
  - ChanRe Rheumatology And Immunology Center And Research, Bangalore, Karnataka
  - Sushruta Multispecialty Hospital & Research Center Pvt Ltd, Hubli, Karnataka
  - Kasturba Medical College Hospital, Mangalore, Madhav Nagar, Manipal, Karnataka
  - Jasleen Hospital, Nagpur, Maharashtra
  - Synexus Affiliate - Sujata Birla Hospital & Medical Research Center, Nashik, Maharashtra
  - Fortis Escorts Hospital, Jaipur, Rajasthan
- Italy (6):
  - Azienda Ospedaliera Universitaria, Modena, MO
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Policlinico Umberto I, Roma
  - Azienda Ospedaliera Santa Maria Della Misericordia, Udine
- Japan (16):
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Jp Red Cross Society Himeji Hp, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - St. Lukes International Hospital, Chuo-Ku, Tokyo
  - Toho University Ohashi Med C, Meguro-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Hamanomachi Hospital, Fukuoka
  - Nippon Medical School Hospital, Tokyo
- Philippines (7):
  - Mary Mediatrix Medical Center, Lipa, Batangas
  - Cebu Doctors Hospital, Cebu City, Cebu
  - Southern Philippines Medical Center, Davao City, Davao Del Norte
  - Angeles University Foundation and Medical Center, Angeles City, Pampanga
  - Chong Hua Medical Arts Center, Cebu City
  - Makati Medical Center, Makati City
  - St. Luke's Medical Center, Quenzon City
- Poland (14):
  - Niepubliczny Zaklad Opieki Zdrowotnej Biogenes Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Medycyna Kliniczna, Warsaw, Masovian Voivodeship
  - Reumatika - Centrum Reumatologii, Warsaw, Masovian Voivodeship
  - Gabinet Internistyczno- Reumatologiczny Piotr Adrian Klimiuk, Bialystok, Podlaskie Voivodeship
  - Zespol Poradni Specjalistycznych REUMED, Lublin, Polska
  - Ambulatorium Barbara Bazela, Elblag, Warminsko-Mazurki
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej, Bydgoszcz
  - Centrum Medyczne Pratia Katowice, Katowice
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Centrum Medyczne Plejady, Krakow
  - NZOZ Lecznica MAK-MED s.c., Nadarzyn
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny UM w Poznaniu, Poznan
  - Centrum Medyczne AMED, Warsaw
- Romania (8):
  - Napoca Emergency Clinical County Hospital, Cluj-Napoca, Cluj
  - Craiova Emergency Clinical County Hospital, Craiova, Dolj
  - SC CMDTA Neomed SRL, Brasov
  - Spitalul Clinic Sf Maria Bucuresti, Bucharest
  - Spitalul Clinic "Dr. Ioan Cantacuzino", Bucharest
  - SANA Medical Center, Bucharest
  - St. Maria Clinical Hospital, Bucharest
  - Spitalul Euroclinic, Bucureti
- Serbia (5):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Institute for Treatment and Rehabilitation Niska Banja, Niška Banja
  - Clinical Center of Vojvodina, Novi Sad
- South Africa (7):
  - Suite 509 Umhlanga Netcare Medical Centre, Umhlanga, Durban
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Guateng
  - Jakaranda Hospital, Muckleneuk, Pretoria
  - Panorama Medical Centre, Cape Town, Western Cape
  - Arthritis Clinical Trial Centre, Pinelands, Western Cape
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
  - University Of Pretoria, Pretoria
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyung Pook National University Hospital, Daegu, Korea
  - Gachon University Gil Hospital, Incheon, Korea
  - Hanyang University Medical Center, Seoul, Korea
  - The Catholic University of Korea-Seoul St. Mary's Hospital, Seocho-Gu, Seoul
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (7):
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Corporacion Sanitaria Parc Tauli, Sabadell, Sapin
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Corporació Sanitària Clínic, Barcelona
  - Hospital Quiron Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Yin J, Hou Y, Wang C, Qin C. Clinical outcomes of baricitinib in patients with systemic lupus erythematosus: Pooled analysis of SLE-BRAVE-I and SLE-BRAVE-II trials. PLoS One. 2025 Apr 30;20(4):e0320179. doi: 10.1371/journal.pone.0320179. eCollection 2025. PMID 40305472
- [Derived] Petri M, Bruce IN, Dorner T, Tanaka Y, Morand EF, Kalunian KC, Cardiel MH, Silk ME, Dickson CL, Meszaros G, Zhang L, Jia B, Zhao Y, McVeigh CJ, Mosca M. Baricitinib for systemic lupus erythematosus: a double-blind, randomised, placebo-controlled, phase 3 trial (SLE-BRAVE-II). Lancet. 2023 Mar 25;401(10381):1011-1019. doi: 10.1016/S0140-6736(22)02546-6. Epub 2023 Feb 24. PMID 36848919
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: A Study of Baricitinib in Participants With Systemic Lupus Erythematosus — https://trials.lillytrialguide.com/en-US/trial/MnvCKtj7wIG0g4Wo2ugIc

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 2 placebo tablets: one placebo tablet matching 4 milligram (mg) baricitinib and one placebo tablet matching 2 mg baricitinib administered orally once daily (QD) for 52 weeks.
- 2 mg Baricitinib: Participants received one 2 mg baricitinib tablet and one placebo tablet matching 4 mg baricitinib administered QD for 52 weeks.
- 4 mg Baricitinib: Participants received one 4 mg baricitinib tablet and one placebo tablet matching 2 mg baricitinib administered QD for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Started | 257 | 262 | 259
Received at Least One Dose of Study Drug | 256 | 261 | 258
Safety Population (All randomized participants who received at least one dose of study drug and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first postbaseline visit.) | 256 | 261 | 258
Pharmacokinetic (PK) Population (Participants with estimated glomerular filtration rate less than (<) 60 milliliter/minute (mL/min)/1.73 square meter (m2) at screening randomized to the 4 mg dose received a dose of 2 mg QD.) | 0 | 277 | 241
Completed | 212 | 222 | 205
Not Completed | 45 | 40 | 54
Not completed — Adverse Event | 15 | 10 | 16
Not completed — Death | 3 | 0 | 4
Not completed — Lack of Efficacy | 4 | 8 | 8
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Withdrawal by Subject | 18 | 14 | 21
Not completed — Withdrawal by Principal Investigator (PI) | 1 | 1 | 1
Not completed — Sponsor's Decision | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Decreased Neutrophils due to Systemic Lupus Erythematosus (SLE) | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Due to Epidemic/Pandemic | 0 | 1 | 0
Not completed — Randomized but Never Treated | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Total
Number analyzed (Participants) | 256 | 261 | 258 | 775
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (13.47) | 42.80 (12.99) | 42.20 (12.11) | 42.80 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 246 | 245 | 732
  Male | 15 | 15 | 13 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 8 | 28
  Not Hispanic or Latino | 40 | 38 | 40 | 118
  Unknown or Not Reported | 207 | 212 | 210 | 629
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 12 | 13 | 39
  Asian | 71 | 66 | 70 | 207
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 17 | 23 | 26 | 66
  White | 145 | 152 | 140 | 437
  More than one race | 5 | 4 | 4 | 13
  Unknown or Not Reported | 4 | 4 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 34 | 29 | 29 | 92
  Chile | 8 | 14 | 12 | 34
  Colombia | 17 | 15 | 16 | 48
  France | 3 | 2 | 2 | 7
  India | 32 | 28 | 34 | 94
  Italy | 2 | 2 | 5 | 9
  Japan | 14 | 12 | 12 | 38
  Philippines | 13 | 14 | 11 | 38
  Poland | 26 | 36 | 31 | 93
  Romania | 12 | 11 | 7 | 30
  Serbia | 15 | 20 | 18 | 53
  South Africa | 14 | 15 | 12 | 41
  South Korea | 4 | 7 | 8 | 19
  Spain | 12 | 6 | 12 | 30
  United States | 50 | 50 | 49 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index 4 (SRI-4) Response (4 mg Baricitinib)
Description: SRI-4 response defined as 1)greater than or equal to (>=) 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score 2)no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score and 3)no worsening in Physician Global Assessment (PGA) of Disease Activity (worsening defined as an increase of >=0.3 from baseline on a 0-3 visual analogue scale).
  SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms,or laboratory parameters related to Systemic Lupus Erythematosus (SLE),divided into 9 organ systems. For each organ system A=severe disease,B=moderate disease,C=mild stable disease,D=inactive,but previously active,E=inactive and never affected. PGA assess disease activity on a visual analogue scale from 0 to 3 (1=mild, 2=moderate, 3=severe).
Time Frame: Week 52
Population: All randomized participants who received at least one dose of study drug (modified intent-to-treat (mITT) population). The hybrid imputation method [nonresponder imputation (NRI) + multiple imputation (MI)] was used to estimate the response rate in percentage and not the number of responder.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 4 mg Baricitinib
Number analyzed (Participants) | 256 | 258
percentage of participants | 45.6 | 47.1
Statistical Analysis 1: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.711, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.75 to 1.53]

2. Secondary Outcome: Percentage of Participants Achieving SRI-4 Response (2 mg Baricitinib)
Description: as for outcome 1
Time Frame: Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population). The hybrid imputation method [nonresponder imputation (NRI) + multiple imputation (MI)] was used to estimate the response rate in percentage and not the number of responder.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib
Number analyzed (Participants) | 256 | 261
percentage of participants | 45.6 | 46.3
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.789, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.73 to 1.50]

3. Secondary Outcome: Percentage of Participants Achieving a Lupus Low Disease Activity State (LLDAS)
Description: The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. The LLDAS response criteria were: (1) SLEDAI-2K <=4, with no activity in major organ systems (CNS, vascular, renal, cardiorespiratory and constitutional); where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0. (2) no new features of lupus disease activity compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0; (3) PGA (scale 0-3), <=1; (4) current prednisolone (or equivalent) dose <=7.5 mg daily.
Time Frame: Week 52
Population: All randomized participants who received at least 1 dose of study drug (mITT population). The hybrid imputation method [nonresponder imputation (NRI) + multiple imputation (MI)] was used to estimate the response rate in percentage and not the number of responder.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 256 | 261 | 258
percentage of participants | 23.2 | 24.0 | 25.4
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.673, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.72 to 1.68]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.528, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.75 to 1.75]

4. Secondary Outcome: Time to First Severe Flare
Description: Time to first severe flare analyzed using a Cox proportional hazards model with treatment group, baseline disease activity [Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) <10; SLEDAI-2K ≥10], baseline corticosteroid dose (<10 mg/day; ≥10 mg/day prednisone or equivalent), and region fitted as explanatory variables. Participants who did not have severe flare during the flare exposure time period were censored at the end of the flare exposure time.
Time Frame: Baseline to Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 256 | 261 | 258
weeks | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached, and 95% confidence interval could not be calculated. | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached, and 95% confidence interval could not be calculated. | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached, and 95% confidence interval could not be calculated.

5. Secondary Outcome: Percentage of Participants Whose Average Prednisone Dose Had Been Reduced by >=25% From Baseline to <=7.5 mg/Day During Weeks 40 Through 52 in Participants Receiving Greater Than 7.5 mg/Day at Baseline
Description: For the analysis of steroid use, steroid dosages were converted to a prednisone equivalent in mg. A responder was defined as having a prednisone reduction by >=25% from Baseline to <=7.5 mg/day during Weeks 40 through 52.
Time Frame: Baseline, Week 40 through Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population) and had received >7.5 mg prednisone at baseline. Missing data was imputed using the hybrid imputation method [NRI + mLOCF (modified last observation carried forward)].
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 104 | 114 | 105
percentage of participants | 31.7 | 29.8 | 34.3
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.761, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.51 to 1.64]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.611, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.65 to 2.10]

6. Secondary Outcome: Change From Baseline in Worst Pain Numeric Rating Scale (NRS)
Description: Participants assessed the worst pain in the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The average worst daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point. Higher score indicated severe pain. Least Squares (LS) mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >= 10 mg/day prednisone or equivalent), region (North America, Central/South, America/Mexico, Europe, Asia Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at the specified time point. Missing data was imputed using the hybrid imputation method (NRI + MMRM).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 183 | 182 | 179
score on a scale | -1.37 (0.14) | -1.45 (0.14) | -1.44 (0.14)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.698, Mixed Models Analysis; LS Mean difference (Final Values) = -0.08, 95% CI 2-sided [-0.47 to 0.32], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.744, Mixed Models Analysis; LS Mean difference (Final Values) = -0.07, 95% CI 2-sided [-0.46 to 0.33], Standard Error of Mean 0.20

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Total Score
Description: FACIT-Fatigue score calculated according to a 13-item questionnaire that assess self reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse possible score) to 52 (best score). A higher score reflected an improvement in the participant's health status. Least Squares (LS) mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >= 10 mg/day prednisone or equivalent), region (North America, Central/South, America/Mexico, Europe, Asia Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 200 | 203 | 193
score on a scale | 7.26 (0.60) | 6.90 (0.60) | 6.96 (0.61)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.665, Mixed Models Analysis; LS Mean difference (Final Values) = -0.36, 95% CI 2-sided [-2.00 to 1.28], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.723, Mixed Models Analysis; LS Mean difference (Final Values) = -0.30, 95% CI 2-sided [-1.95 to 1.35], Standard Error of Mean 0.84

8. Secondary Outcome: Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Total Activity Score ≥10 at Baseline With ≥50% Reduction in CLASI Total Activity Score
Description: The CLASI is a single-page tool that separately quantifies disease activity and damage. For the activity score, points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
Time Frame: Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population) and had baseline CLASI score >=10. Missing data was imputed using NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 59 | 51 | 50
percentage of participants | 66.1 | 56.9 | 58.0
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.372, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.31 to 1.55]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.555, Regression, Logistic; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.34 to 1.78]

9. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: The number of tender and painful joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as tender or not tender. LS mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: tender joint count
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 200 | 201 | 190
tender joint count | -6.92 (0.301) | -7.40 (0.300) | -7.83 (0.306)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.251, Mixed Models Analysis; LS Mean difference (Final Values) = -0.48, 95% CI 2-sided [-1.31 to 0.34], Standard Error of Mean 0.422
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.333, Mixed Models Analysis; LS Mean difference (Final Values) = -0.91, 95% CI 2-sided [-1.74 to -0.07], Standard Error of Mean 0.425

10. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: The number of swollen joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as swollen or not swollen. LS mean was calculated using MMRM analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: swollen joint count
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 200 | 201 | 190
swollen joint count | -4.79 (0.202) | -5.10 (0.201) | -5.31 (0.205)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.284, Mixed Models Analysis; LS Mean difference (Final Values) = -0.30, 95% CI 2-sided [-0.86 to 0.25], Standard Error of Mean 0.282
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.069, Mixed Models Analysis; LS Mean difference (Final Values) = -0.52, 95% CI 2-sided [-1.08 to 0.04], Standard Error of Mean 0.284

11. Secondary Outcome: Population Pharmacokinetics (PK): Area Under the Concentration-Time Curve for Dosing Interval of Baricitinib at Steady State (AUCtau,ss)
Description: AUCtau,ss reported for participants who received multiple doses of mg baricitinib was derived by a population pharmacokinetics approach.
Time Frame: Week 0 (Baseline): 15 minutes (min) and 60 min postdose; Week 4: 2 to 4 hours (hr) postdose; Week 8: 4 to 6 hr postdose; Week 12 and Week 16 predose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 277 | 241
nanogram*hour/milliliter (ng*h/mL) | 257 (48) | 505 (50)

12. Secondary Outcome: Population PK: Maximum Observed Drug Concentration at Steady State (Cmax,ss)
Description: PK: Maximum Concentration of Baricitinib at steady-state (Cmax,ss) was derived by a population pharmacokinetics approach.
Time Frame: as for outcome 11
Population: All randomized participants who received at least one dose of study drug with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 277 | 241
nanograms per milliliter (ng/mL) | 27.0 (23) | 54.1 (24)

ADVERSE EVENTS:
Time Frame: Baseline through Follow-up (Up to 56 Weeks)
Description: All randomized participants who received at least one dose of study drug and who did not discontinue from the study for the reason 'Lost to Follow-up' at the first postbaseline visit (safety population). Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 3/256 | 0/261 | 4/258
Serious Adverse Events (participants affected / at risk) | 26/256 | 35/261 | 32/258
Other Adverse Events (participants affected / at risk) | 96/256 | 100/261 | 96/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=256) | 2 mg Baricitinib (N=261) | 4 mg Baricitinib (N=258)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Disseminated varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster meningomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0/241 (0) | 1/246 (1) | 0/245 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/241 (0) | 1/246 (1) | 0/245 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/241 (1) | 1/246 (1) | 1/245 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/241 (0) | 1/246 (1) | 0/245 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1/241 (1) | 0/246 (0) | 0/245 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=256) | 2 mg Baricitinib (N=261) | 4 mg Baricitinib (N=258)
Neutropenia (Blood and lymphatic system disorders) | 7 (9) | 5 (6) | 13 (19)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 20 (25) | 10 (11)
Nasopharyngitis (Infections and infestations) | 23 (28) | 18 (20) | 21 (27)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 17 (18) | 19 (22)
Urinary tract infection (Infections and infestations) | 26 (32) | 29 (36) | 19 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8) | 15 (20)
Headache (Nervous system disorders) | 23 (26) | 25 (28) | 19 (21)
Hypertension (Vascular disorders) | 9 (9) | 12 (13) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03616964/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03616964/SAP_001.pdf